CLINICAL TRIAL: NCT02914678
Title: Is There an Ideal Dose of Intravenous Fentanyl in the Prehospital Setting: A Prospective Cluster-randomized Comparison of 2 vs. 3 μg/kg/Transport
Brief Title: Is There an Ideal Dose of Intravenous Fentanyl in the Prehospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-PHA2V3
Record Dates: First submitted 2016-09-12; First posted 2016-09-26 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Acute Pain
Keywords: Emergency Medical Services; Analgesics
MeSH Terms: conditions — Acute Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Existing treatment (No Intervention): Business as usual: Ambulance personnel use existing treatment approach (a total of 2 μg/kg fentanyl per transport)
- More liberal treatment (Experimental): Ambulance personnel use a more liberal treatment approach (a total of 3 μg/kg fentanyl per transport)
  Interventions: Other: Fentanyl

INTERVENTIONS:
Other: Fentanyl — Change in protocol from 2 to a total of 3 μg/kg fentanyl per transport
  Arms: More liberal treatment

SUMMARY:
In a previous study the investigators evaluated the apparent efficacy and safety of intravenous fentanyl administered by ambulance personnel and found that 58.4% (CI 56.4-60.4) out of 2348 prehospital patients treated with fentanyl still experienced moderate to severe pain [numeric rating scale (NRS, 0-10) > 3] at hospital arrival. The number of patients with possible fentanyl-related side effects was low.

Therefore, the aim of the present study is to explore the efficacy and safety of a liberalized pain treatment protocol for ambulance personnel (a total of 3 μg/kg per transport) compared with existing restrictive protocol (a total of 2 μg/kg per transport). The investigators hypothesize that:

* A higher proportion of patients will experience sufficient pain relief at hospital admission (NRS < 4) using the liberalized protocol and
* There will be no differences in the proportion of potential fentanyl related side-effects are observed.

DETAILED DESCRIPTION:
A prospective cluster-randomized trial observing proportional differences in sufficient pain relief at hospital admission (NRS < 4) and potential fentanyl related side-effects between patients treated by ambulance personnel applying either:

* a more liberal treatment approach (a total of 3 μg/kg per transport) or
* existing treatment approach (a total of 2 μg/kg per transport).

The Ambulance stations and their affiliated ambulance personnel are stratified into 5 clusters according to size/average transports per month and randomized to either liberal or existing treatment approach within each cluster. As patients are not randomized on an individual level baseline differences between the two groups and its patients are adjusted statistically with relevant confounders on 3 overall levels:

1. Patients: Charlson Comorbidity Index Score, main overall diagnose category, inhospital surrogate measures of disease severity (intensive care unit admission and 30-day mortality).
2. Ambulance personnel: Years of experience and preinterventional cumulative fentanyl administration and
3. Ambulance stations and geographical factors: prehospital time measures and geographical distance from site of emergency to hospital.

These covariates are obtained from the Danish National Patient Registry, the Danish Civil Registration System and the electronic prehospital patient journal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pain treated with intravenous fentanyl by ambulance personnel

Exclusion Criteria:

* Reduced conscious level (GCS < 15) before initiation of fentanyl treatment
* Reduced respiratory rate (< 10/minute) before initiation of fentanyl treatment
* Patient weight < 30 kg
* Known opioid allergy
* Women in labour
* Chronic pain conditions

Max Age: 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7093 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with sufficient pain relief (NRS < 4) at hospital arrival | Up to 6 hours

SECONDARY OUTCOMES:
Proportion of patients with reduced Glasgow Coma Scale (<15) after fentanyl administration and at any given point during transport | Up to 6 hours
Proportion of patients with reduced respiratory rate (<10/minute) after fentanyl administration and at any given point during transport | Up to 6 hours
Proportion of patients with reduced peripheral oxygen saturation (< 90%) after fentanyl administration and at any given point during transport | Up to 6 hours
Proportion of patients with hypotension after fentanyl administration and at any given point during transport | Up to 6 hours
  Hypotension defined as a drop in mean arterial pressure (MAP) >= 10 mmHg to a MAP < 70 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Friesgaard, MD, PhD Student, Principal Investigator — University of Aarhus; Lone Nikolajsen, DmSc, Study Chair — Aarhus University Hospital; Hans Kirkegaard, Professor, Study Chair — Aarhus University Hospital; Erika Frischknecht Christensen, Professor, Study Chair — North Denmark Region; Matthias Giebner, MD, Study Chair — Central Denmark Region; Claus-Henrik Rasmussen, MD, Study Chair — Central Denmark Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friesgaard KD, Nikolajsen L, Giebner M, Rasmussen CH, Riddervold IS, Kirkegaard H, Christensen EF. Efficacy and safety of intravenous fentanyl administered by ambulance personnel. Acta Anaesthesiol Scand. 2016 Apr;60(4):537-43. doi: 10.1111/aas.12662. Epub 2015 Nov 27. PMID 26612100
- [Background] Lynge E, Sandegaard JL, Rebolj M. The Danish National Patient Register. Scand J Public Health. 2011 Jul;39(7 Suppl):30-3. doi: 10.1177/1403494811401482. PMID 21775347
- [Background] Schmidt M, Pedersen L, Sorensen HT. The Danish Civil Registration System as a tool in epidemiology. Eur J Epidemiol. 2014 Aug;29(8):541-9. doi: 10.1007/s10654-014-9930-3. Epub 2014 Jun 26. PMID 24965263
- [Derived] Friesgaard KD, Kirkegaard H, Rasmussen CH, Giebner M, Christensen EF, Nikolajsen L. Prehospital intravenous fentanyl administered by ambulance personnel: a cluster-randomised comparison of two treatment protocols. Scand J Trauma Resusc Emerg Med. 2019 Feb 7;27(1):11. doi: 10.1186/s13049-019-0588-4. PMID 30732618